CLINICAL TRIAL: NCT02357641
Title: Analysis of Myocardial Deformation in Patients With Acute Coronary Disease
Brief Title: Acute Coronary Disease (ACS)- Strain
Acronym: ACS-Strain
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A 13-089
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Cardiac and Non Cardiac Thoracal Disorder
Keywords: acute coronary disease, echographic strain analysis, cut off

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with thoracal disorder: 300 patients with thoracal disorder, cardiac or non- cardiac, are enrolled prospectively to undergo routinely examinations such as clinical and hemodynamic chemistry as well as echocardiography for strain analysis refering to myocardial deformation.
  Especially analysis of strain data (circumferential and radial), regional and global left and right ventricular wall movement data and diastolic parameters will be analysed retrospectively to investigate a probable cut off value corresponding to acute coronary disease or non cardiac disorder (Intervention: retrospective echographic myocardial strain analysis refering to acute coronary syndrome).
  Interventions: Other: retrospective echographic myocardial strain analysis refering to acute coronary syndrome

INTERVENTIONS:
Other: retrospective echographic myocardial strain analysis refering to acute coronary syndrome — retrospective evaluation for cut off value of circumferential and radial echographic strain parameters corresponding to acute coronary disease

SUMMARY:
Examination of probable distinction between cardiac or non- cardiac thoracal disorder via echocardiographic myocardial strain analysis

DETAILED DESCRIPTION:
Patients with cardiac disorder have to undergo time- consuming and expensive examinations such as laboratory of cardiac biomarkers or ischemic diagnostic. To save time and money in this observational registry the probable distinction between cardiac and non- cardiac disorder in patients with vague thoracal disorder and the probability for coronary artery disease (determined via Grace Score) is examined via echographic myocardial strain analysis in 300 patients retrospectively to establish a cut off value corresponding to acute coronary disease also to prevent coronary angiography. Therefore patients undergo echography routinely with consecutive evaluation of systolic, diastolic and strain analysis to elevate exact statements with reference to deformation of the myocard and its velocity. Several study have shown that these strain parameters (circumferential and radial strain) enable vitality and ischemic diagnosis and therefore could be eligible for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* thoracal cardiac or non cardiac disorder
* signed informed consent

Exclusion Criteria:

* glomerular filtration rate (GFR) < 60 ml/min
* angina pectoris
* acute myocardial infarction within 3 months prior inclusion
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with vague thoracal disorder -cardiac or non cardiac- are enrolled prospectively to undergo routinely echography as well as routine examinations such as anamnetic, hemodynamic examinations and laboratory. The distinction between non cardiac disorder or acute coronary disease (ACS) is offen difficult so that time- consuming and expensive ischemic diagnostics or coronary artery angiography will follow. To prevent these time consuming or expensive diagnostics retrospectively a cut off value will be determined of systolic, diastolic and additionally of circumferential and radial echographic strain data analysis corresponding to acute coronary disease.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Determination of cut off value of circumferential and radial myocardial echographic strain data corresponding to acute coronary disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schroeder, MD, Principal Investigator — University Hospital Aachen, Clinic of Cardiology, Angiology, Pneumology and Intensive Care Medicine
Locations (1):
- Department of Cardiology, RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Schroeder J, Hamada S, Grundlinger N, Rubeau T, Altiok E, Ulbrich K, Keszei A, Marx N, Becker M. Myocardial deformation by strain echocardiography identifies patients with acute coronary syndrome and non-diagnostic ECG presenting in a chest pain unit: a prospective study of diagnostic accuracy. Clin Res Cardiol. 2016 Mar;105(3):248-56. doi: 10.1007/s00392-015-0916-2. Epub 2015 Sep 8. PMID 26349786